CLINICAL TRIAL: NCT01368185
Title: A Retrospective Survey to Evaluate the Impact of Hyzaar on Uric Acid in the Management of Hypertensive Patients in Normal Practice
Brief Title: Impact of MK-0954A on Uric Acid in the Management of Hypertension (MK-0954A-366)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0954A-366; MK-0954A-366
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Results first posted 2011-09-01 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Essential hypertension Uric acid Retrospective Hyzaar
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants with hypertension who had been treated with MK-0954A (losartan potassium 50 mg + hydrochlorothiazide 12.5 mg) for at least three months

SUMMARY:
This was a retrospective, chart review, observational study to assess the effect of MK-0954A (losartan potassium 50 mg + hydrochlorothiazide 12.5 mg [Hyzaar(R)]) treatment for a period of at least three months on serum uric acid levels.

ELIGIBILITY:
Inclusion criteria:

* Participant was >20 years and <75 years of age on the index date (i.e., the date of initiating MK-0954A therapy)
* Diagnosed with hypertension and had received MK-0954A 50/12.5 mg for at least 3 months
* Had at least one serum uric acid measurements at baseline and one at 3 months after using MK-0954A 50/12.5 mg
* Had the following records documented in the chart during the data collection period:

  * medical history and co-morbidities (if available)
  * sitting blood pressure, serum uric acid, lipid profile test results before and after using MK-0954A 50/12.5 mg
  * serum electrolytes, serum creatinine, and pre-meal sugar (if available)
  * prescription information of all antihypertensive regimens

Exclusion criteria:

* Had been treated with diuretic or angiotensin-receptor blockers (ARBs) 2 weeks before initiated treatment with MK-0954A 50/12.5 mg
* Serum creatinine >2 mg/dL

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from 33 physicians from different levels of hospitals were invited to provide information on patients who received MK-0954A and had pre- and post-treatment serum uric acid and lipid profile reports during the study period. Each physician could provide up to 30 clinical charts of patients matching the inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1705 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the medical charts of the eligible study patients were reviewed. The study index period (when patients had to have received treatment for 3 months) was from June 1st 2007 to December 31st 2008. Data were collected retrospectively between November 2008 and August 2010.
Pre-assignment Details: 1735 patients were enrolled into this study. Among them, 1705 patients were eligible after excluding 30 patients.
Period: Overall Study
Arm/Group | All Participants
Started | 1705
Completed | 1705
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1705
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 795
  Male | 910

OUTCOME MEASURES:

1. Primary Outcome: Serum Uric Acid (SUA) Level
Description: SUA at baseline and Month 3.
Time Frame: Baseline and Month 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 1705
mg/dL
  Baseline | 6.4 (1.6)
  Month 3 | 6.6 (1.6)
Statistical Analysis 1: Comparison: All Participants; Comparison between Month 3 and Baseline; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; % change SUA from baseline = 4.6, Standard Deviation 0.9 — Percent change of month 3 SUA minus baseline SUA

2. Secondary Outcome: The Percentage of Patients With Hyperuricemia
Description: Hyperuricemia was defined as SUA >6.6mg/dL in females and >7.7mg/dL in males.
Time Frame: Baseline and Month 3
Measure: Number; unit: percent of participants
Arm/Group | All Participants
Number analyzed (Participants) | 1705
percent of participants
  Baseline | 27.0
  Month 3 | 14.6
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < 0.0001, McNemar

3. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: DBP at baseline and month 3.
Time Frame: Baseline and Month 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 1705
mmHg
  Baseline | 89 (13)
  Month 3 | 81 (9)
Statistical Analysis 1: Comparison: All Participants; Comparison between Month 3 and Baseline; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; % change DBP from Baseline = -7.1, Standard Deviation 0.4 — Percent change of month 3 DBP minus baseline DBP (n=1239)

4. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: SBP at baseline and month 3.
Time Frame: Baseline and Month 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 1705
mmHg
  Baseline | 150 (19)
  Month 3 | 135 (15)
Statistical Analysis 1: Comparison: All Participants; Comparison between Month 3 and Baseline; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; % change SBP from Baseline = -9.1, Standard Deviation 0.3 — Percent change of month 3 SBP minus baseline SBP (n=1245)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/1705
Other Adverse Events (participants affected / at risk) | 7/1705
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1705)
Dizziness (Nervous system disorders) | 3 (3)
Tachycardia/Palpitation (Cardiac disorders) | 2 (2)
Dyspnea with wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mild cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.